CLINICAL TRIAL: NCT02350270
Title: Gait, cOgnitiOn & Decline (GOOD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Biomathics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2014-17
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2014-02

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Moderate Dementia; Healthy
Keywords: cognitively healthy individuals
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Gait; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- cognitively healthy individuals (CHI): CHI were participants without objective cognitive impairment
  Interventions: Other: gait and cognitive testing
- mild cognitive impairment (MCI): MCI was diagnosed if participants met the following criteria: presence of spontaneous cognitive complaints and objective cognitive impairment
  Interventions: Other: gait and cognitive testing
- mild and moderate dementia: Diagnoses of dementia were assigned according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV TR, 2000; Association, 2000; 22) at consensus diagnostic case conferences
  Interventions: Other: gait and cognitive testing

INTERVENTIONS:
Other: gait and cognitive testing

SUMMARY:
The main objective of the GOOD initiative was to determine which spatio-temporal gait parameters and/or combination(s) of spatio-temporal gait parameters best differentiate between cognitively healthy individuals (CHI), patients with mild cognitive impairment (MCI) and those with mild and moderate dementia.

DETAILED DESCRIPTION:
Gait disorders are frequent in individuals with cognitive disorders. However, the profile of spatio-temporal gait parameters in the different cognitive status in aging (from normal cognition to dementia) has been poorly studied. Determining this profile associated with the severity of cognitive disorders may be helpful to understand the complex interplay between gait and cognitive disorders and, thus, may have important implication for the diagnosis process of patients with and without dementia. For instance, defining a motor phenotype of the severity of cognitive disorders by using quantitative gait measurements could be used to improve the prediction and the diagnosis of dementia.

The investigators hypothesized that, compared to CHI, people with MCI and mild dementia could be characterized by specific phenotypes of spatio-temporal gait parameters measured with the GAITRite® system, and that these profiles could be explained by declines in domain-specific cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Being 60 years old and older
* Ability to answer questions

Exclusion Criteria:

* Opposition to the use of information collected for research purposes

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were recruited in each memory clinic by a physician
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Spatio-temporal gait parameters | This outcome is assessed at inclusion
  Spatio-temporal gait parameters were measured at steady state walking using GAITRite®-system.

SECONDARY OUTCOMES:
Clinical assessment | This outcome is assessed at inclusion
  This outcome was assessed by a questionnaire.
Cognitive status | This outcome is assessed at inclusion
  Cognitive status was assessed by cognitive testing.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- University Hospital, Angers, France